CLINICAL TRIAL: NCT02998489
Title: Effectiveness and Safety of Rapid Enteral Feeding in Preterm Infants Between 1000 and 2000 Grams of Birth Weight
Brief Title: Effectiveness and Safety of Fast Enteral Feeding in Preterm Infants Between 1000 and 2000 Grams of Birth Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/25
Record Dates: First submitted 2016-12-11; First posted 2016-12-20 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Feeding Behavior
Keywords: enteral nutrition; infant,premature; feeding method
MeSH Terms: conditions — Feeding Behavior; Premature Birth | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fast milk advancement (Experimental): 30-40 cc/kg/d of human milk or formula milk administered by orogastric tube or by suction
  Interventions: Other: Fast milk advancement
- Traditional milk advancement (Active Comparator): 20 cc/kg/d of human milk or formula milk administered by orogastric tube or by suction
  Interventions: Other: Traditional milk advancement

INTERVENTIONS:
Other: Fast milk advancement — 30-40 cc/kg/d of human milk or formula milk until total enteral feeding has been achieved
  Other Names: Milk
  Arms: Fast milk advancement
Other: Traditional milk advancement — 20 cc/kg/d of human milk or formula milk until total enteral feeding has been achieved
  Other Names: Milk
  Arms: Traditional milk advancement

SUMMARY:
This is a randomized controlled trial with infants less than 34 weeks and between 1000 and 2000 grams at birth, that seeks to establish the safety and effectiveness of fast enteral advancement (milk 30-40 cc/kg/d) compared with traditional advancement (milk 20 cc/kg/d)

DETAILED DESCRIPTION:
Progression of enteral feeding in preterm infants is still controversial. The neonatologist needs to provide adequate caloric intake avoiding the risk of food intolerance and necrotizing enterocolitis.

Objective: To establish the safety and effectiveness of fast enteral advancement compared with traditional advancement.

Design: A randomized controlled clinical trial with infants less than 34 weeks and between 1000 and 2000 grams at birth conducted at Hospital Universitario San Ignacio in Bogotá, Colombia.

Methods: 30 cc versus 20 cc / kg / day advancing in infants between 1000 and 1499g and 40cc versus 20 cc / kg / day advancing in infants between 1500 and 1999g.

Outcomes: days to reach full enteral nutrition, days of parenteral nutrition (PN) and/or intravenous fluids (IVF), days to regain birth weight, episodes of food intolerance, anthropometric measurements and weight gain at 40 weeks; rate of late onset sepsis, hypoglycemia, hyperbilirubinemia, necrotizing enterocolitis (NEC) and mortality. Data will be analyzed with Student t test or Mann-Whitney U-test and Pearson Chi-square or Fisher test. Multiple linear regression will be performed.

Ethics: This Protocol was approved by the Ethics and Research Committee of Pontificia Universidad Javeriana and San Ignacio Hospital. Informed consent will be requested to parents.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 34 weeks of gestational age.
* Weight at birth between 1000 and 2000 grams.
* Infants hospitalized in the newborn unit at Hospital Universitario San Ignacio in Bogotá, Colombia.

Exclusion Criteria:

* Perinatal Asphyxia
* Intrauterine Growth Restriction
* Diagnosis of Congenital Hearth Disease
* Severe Hypoxemia
* Major Congenital Malformations
* Metabolic Disease
* Intolerance to initiate oral feeding at the eligibility
* Patent Ductus with hemodynamic instability
* Early Onset Sepsis with hemodynamic instability
* Refusal of parents to participate in the study

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
days to reach full enteral nutrition | number of days from date of randomization until the day that the baby reach full enteral nutrition or date of death from any cause assessed up to 12 weeks
  number of days employed to reach full enteral nutrition with breast milk, formula milk or breast milk plus formula milk.
days of intravenous fluids | number of days of intravenous fluids from birth until suspension of them or date of death from any cause assessed up to 12 weeks
  number of days with intravenous fluids included parenteral nutrition and dextrose with electrolytes

SECONDARY OUTCOMES:
days to regain birth weight | number of days from birth, employed to regain birth weight or date of death from any cause assessed up to 12 weeks
  number of days employed to regain birth weight
episodes of food intolerance | number of episodes of food intolerance per day from date of randomization until hospital discharge or date of death from any cause assessed up to 12 weeks
  number of episodes of food intolerance per day during hospitalization
weight at 40 weeks | weight at 40 weeks of post menstrual age
  weight in grams at 40 weeks of post menstrual age
length at 40 weeks | length at 40 weeks of post menstrual age
  length in centimeters at 40 weeks of post menstrual age
head circumference at 40 weeks | head circumference at 40 weeks of post menstrual age
  head circumference in centimeters at 40 weeks of post menstrual age
weight gain per day at 40 weeks of post menstrual age | weight gain in grams per day from birth until 40 weeks of post menstrual age
  weight gain in gr./d from birth until 40 weeks of post menstrual age
rate of necrotizing enterocolitis | through study completion(from date of randomization until 40 weeks of post menstrual age)
  rate of necrotizing enterocolitis through study completion
rate of mortality | through study completion(from date of randomization until 40 weeks of post menstrual age)
  number of patients who died during the study's follow up
rate of late onset sepsis | from date of randomization until hospital discharge or date of death from any cause assessed up to 12 weeks
  number of patients who had late onset sepsis during hospitalization
rate of hyperbilirubinemia | from date of randomization until hospital discharge or date of death from any cause assessed up to 12 weeks
  number of patients who had hyperbilirubinemia and were treated with phototherapy during hospitalization
rate of hypoglycemia | from date of randomization until hospital discharge or date of death from any cause assessed up to 12 weeks
  number of patients who had hypoglycemia during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Montealegre, Dr., Principal Investigator — Hospital Universitario San Ignacio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morgan J, Young L, McGuire W. Slow advancement of enteral feed volumes to prevent necrotising enterocolitis in very low birth weight infants. Cochrane Database Syst Rev. 2015 Oct 15;(10):CD001241. doi: 10.1002/14651858.CD001241.pub6. PMID 26469124
- [Result] Moore TA, Wilson ME. Feeding intolerance: a concept analysis. Adv Neonatal Care. 2011 Jun;11(3):149-54. doi: 10.1097/ANC.0b013e31821ba28e. PMID 21730906